CLINICAL TRIAL: NCT02117752
Title: Dermal Tolerability of Dapsone Gel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 225678-009
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sodium Dodecyl Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapsone Gel Subset 1 (Experimental): Dapsone gel, dapsone gel vehicle and controls applied to the skin by separate occlusive patches every 24 hours for 21 days followed by a 10 to 17 day rest period then one application each of dapsone gel and dapsone gel vehicle by patch for 48-hours.
  Interventions: Drug: dapsone gel; Drug: dapsone gel vehicle; Drug: sodium lauryl sulfate; Drug: Normal saline
- Dapsone Gel Subset 2 (Experimental): Dapsone gel, dapsone gel vehicle and negative control applied to the skin by separate occlusive patches every 48 to 72 hours for 21 days followed by a 10 to 17 day rest period then one application each of dapsone gel and dapsone gel vehicle by patch for 48-hours.
  Interventions: Drug: dapsone gel; Drug: dapsone gel vehicle; Drug: Normal saline

INTERVENTIONS:
Drug: dapsone gel — Patches containing dapsone gel will be applied to the skin.
Drug: dapsone gel vehicle — Patches containing dapsone gel vehicle will be applied to the skin.
Drug: sodium lauryl sulfate — Patches containing sodium lauryl sulfate (Positive Control) will be applied to the skin.
  Arms: Dapsone Gel Subset 1
Drug: Normal saline — Patches containing normal saline (Negative Control) will be applied to the skin.

SUMMARY:
This study will determine the cumulative irritation potential and sensitization potential of dapsone gel and vehicle after repeat applications on the skin of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

-Healthy adults.

Exclusion Criteria:

* Skin diseases, excessive hair, tattoos, pigmentation, scars or moles that could interfere with patch application
* Sensitivity to adhesive bandages or tape.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mean Cumulative Irritation Index During Induction Phase | 21 Days
Incidence of Sensitization Reactions During Challenge Phase | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fair Lawn, New Jersey, United States